CLINICAL TRIAL: NCT05402553
Title: The Efficacy of Adjunctive Use of Ondansetron in Patients With Sepsis and Septic Shock
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Noha Mansour (Other)
Responsible Party: Sponsor-Investigator, Noha Mansour, Principal investigator-Lecturer of Clinical Pharmacy-Clinical Pharmacy and Pharmacy Practice Department, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-2022
Record Dates: First submitted 2022-05-30; First posted 2022-06-02 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator)
  Interventions: Drug: Ondansetron
- Control (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ondansetron — patients will receive, in addition to standard therapy, ondansetron IV bolus 8 mg BID for 3 days
  Arms: Intervention
Drug: Placebo — patients will receive, in addition to standard therapy, normal saline IV bolus BID for 3 days
  Arms: Control

SUMMARY:
Sepsis is a systemic inflammatory response that has deleterious effects and considered the leading cause of death in critically ill patients 1 . One of the hallmarks of severe sepsis is the progressive, injurious inflammatory response to infection, mediated by the excessive release of inflammatory mediators and consequently, associated with multiple organs damage 2 . Various studies have demonstrated that adverse outcomes in sepsis patients are closely related to the development of myocardial dysfunction 3 . The mortality of sepsis combined with cardiac functional insufficiency has increased significantly to 70%-90% 4 . Therefore, targeting cardiac insufficiency and heart injury may represent a novel treatment strategy. Several reports documented critical involvement of serotonin 5-hydroxytryptamine in the pathogenesis of sepsis. The aim of the current study is to evaluate the efficacy of ondansetron adjuvant use in patients with sepsis and septic shock.

ELIGIBILITY:
Inclusion Criteria:

male or female adult patients, aged 18 years or older with sepsis or septic shock after surgery according to the 2016 third international consensus definitions for sepsis and septic shock

Exclusion Criteria:

diagnosis of septic shock longer than 24 hours ago known or suspected disease with a strong indication or contraindication for the study drugs Pregnant and lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04-24 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Sequential organ failure assessment (SOFA score) | 3 days post randomization
  Difference between study groups in mean change from baseline in SOFA score

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided